CLINICAL TRIAL: NCT01480349
Title: Shunt Outcomes of Post-Hemorrhagic Hydrocephalus: A Network Pilot Study
Brief Title: Shunt Outcomes of Post-Hemorrhagic Hydrocephalus
Acronym: SOPHH
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 46249; 1RC1NS068943-01 (NIH); HCRN 005 (Other: HCRN Protocol Number)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Post-Hemorrhagic Hydrocephalus
Keywords: Post-Hemorrhagic Hydrocephalus; Intraventricular Hemorrhage; Low Birth Weight Premature Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter, prospective pilot study will compare the effectiveness of two established procedures used in the treatment of post-hemorrhagic hydrocephalus in very low birth weight infants, specifically ventricular reservoirs and subgaleal shunts. The study is being conducted by the Hydrocephalus Clinical Research Network (HCRN), a network established to conduct multi-institutional clinical trials on pediatric hydrocephalus.

DETAILED DESCRIPTION:
Intraventricular hemorrhage and post-hemorrhagic hydrocephalus remain a leading cause of mortality and long-term morbidity in premature infants. The two most common temporary cerebrospinal fluid (CSF) diversion procedures are the ventriculosubgaleal shunt (SGS) and an implanted ventricular reservoir (RES) for intermittent CSF removal. These methods are physiologically very different and their comparative effectiveness in treating hydrocephalus and possibly reducing the need for an eventual permanent CSF shunt is currently not known. The goal of this pilot study is to obtain information critical for planning and executing a future randomized trial comparing SGS and RES. Specifically, this pilot study will establish inclusion criteria, define the primary outcome, and standardize the interventions in preparation for initiating a comparative trial between the SGS and RES procedures. In addition, the importance of examining the neurodevelopmental outcomes for these patients has been recognized within the neurosurgical and neuropsychological settings. Therefore, the scope of this study has been extended to include an examination of the neurodevelopmental outcomes at 18 to 22 months and at 36 to 42 months in patients who undergo BSID-III testing at their clinical centers.

ELIGIBILITY:
Inclusion Criteria:

* premature neonates with birth weights less than 1500 grams
* Grade III or IV intraventricular hemorrhage
* Fronto-occipital horn ratio greater than or equal to 0.50

Exclusion Criteria:

* Less than 72 hour life expectancy from other medical problems

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All premature neonates with grade III or IV intraventricular hemorrhage who primarily present or are referred prior to surgical intervention for post hemorrhagic hydrocephalus to HCRN Clinical Centers.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
Specific Aim I: Proportion of temporization | 5 years
  The proportion of all infants entering the study who meet the criteria for surgical temporization.
Specific Aim 2: Conversion proportion | 5 years
  The proportion of all infants with SGS or RES who met criteria for conversion to permanent shunt.
Specific Aim 3: Surgery Checklist Scores | 5 years
  Surgery checklist scores of individual surgeon performance in standardized procedures.

SECONDARY OUTCOMES:
Protocol adherence | 5 years
  Protocol adherence by network, center, surgeon, decision rubric, and individual decision data points.
CSF Infection | 5 years
  Incidence of CSF infection while on the protocol.
Neurodevelopmental Outcomes | 7 years
  Subscores from the Bayley Scales of Infant Development, version III (BSID-III) to include cognitive, language and motor subtests will be obtained for patients undergoing BSID-III testing at 18-22 and 36-42 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: John C Wellons, III, MD, Study Chair — Vanderbilt University Medical Center; Chevis N Shannon, MBA, DrPH, Principal Investigator — Vanderbilt University Medical Center
Locations (7):
- United States (6):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Sick Children's Hospital, Toronto, Ontario, Canada

REFERENCES:
- See also: Hydrocephalus Clinical Research Network website — http://hcrn.org